CLINICAL TRIAL: NCT05496621
Title: Validity and Reliability of Turkish Version of Keele STarT MSK Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yasemin Çırak, Professor, Istinye University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 003
Record Dates: First submitted 2022-02-07; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Musculoskeletal Diseases
Keywords: musculoskeletal diseases
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Our work will be carried out in two stages. 1st stage Keele start msk tool translated into Turkish and its cultural adaptation, 2nd stage statistical analysis of the reliability and validity of the Turkish Keele start msk tool. Permission was obtained from Keele University, the developer of the scale, before starting the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Musculoskeletal Diseas (Experimental): Questionnaires will be asked for the validity of the Turkish version of the Keel Start Tool.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — 1st Stage Keele Start MSk tool translated into Turkish and its cultural adaptation, 2nd Stage Statistical analysis of reliability and validity of Turkish Keele start msk tool

SUMMARY:
The aim of this study is to investigate the usability of the Turkish version of the Keel Start Tool as a valid and reliable method in groups with 5 different types of musculoskeletal pain (knee, neck, shoulder, back, multiple painful areas). When the literature is examined, Turkish validity has not been made in this area.

DETAILED DESCRIPTION:
SK diseases are the 3 most common disease groups in Turkey, and it has been determined that the rate of discomfort in Turkey is 99%. Although MSK diseases are mostly caused by occupational problems in Turkey, there are clearly information losses and deficiencies in cases such as the risk factors of employers and employees, occupational therapy, lack of insurance payments due to job loss. The study was conducted with 582 office workers. As a result of the study, it was revealed that 55.1% of the participants had back pain and 5% of the participants had back pain, and the rate of women in low back pain was higher.

Keel Start MSK Tool is a tool that provides patients with an appropriate treatment approach, minimizes harm and maximizes treatment benefit. Keele Start MSK Tool msk has been successfully developed for primary care in patients, and it categorizes patients by scoring 9 items and categorizing them into subgroups. This tool is a validated prognostic tool (Keele STarT MSK) with established cut-off points to stratify patients with the five most common musculoskeletal (back, neck, knee, shoulder, multiple painful areas) pain into low, intermediate, and high-risk subgroups. provides 108 patients with low back pain were included in the French version of the Keele STarT Low Back Screening Tool (SBST).

In the UK, which started in 2014, with 1200 patients on MSC pain, stratified; No significant change was achieved as a result of this study, which aims to investigate clinical and cost-effectiveness, as well as to reduce clinician's treatment variability and improve patient outcomes (quality of life, physical function, etc.) since the study has not been completed yet.

In another study, general practitioners screened 3063 patients (1591 interventions, 1472 controls). The EMR template included 1237 eligible patients (513 interventions, 724 controls), while 524 consented to data collection (231 interventions, 293 controls). Although the target of participation was 12 weeks, it took 28 weeks. The target for follow-up was 75% and above and a follow-up rate of over 90% was achieved. As a result of this study, the applicability of the randomized controlled trial design was found to be successful. In addition, the accuracy rate of matched treatment options was also high.

In another UK study, 8 general examinations were randomized (4' stratified care, 4 as regular care) and patients had CNS pain in one of the 5 most common sites. A baseline questionnaire was obtained from the patients, and >90% of these 524 patients were followed up for 8 months. Audio recording or video was taken during the examination. Some patients stated that they wanted to clarify the questions asked, but they could not express themselves well because they had to answer only "yes" or "no" because of this scale. The opinion of the doctors, on the other hand, stated that the result of the Keel Start MSK Tool scale and the treatment approach provided them clinically guiding and different perspectives.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be 18 years or older.
* The location of MSC pain must be one of the 5 regions. These 5 regions; knee, shoulder, back, neck, multi-region.
* Volunteering to participate in the study
* The patient's pain must be chronic. chronic pain; If there is general agreement on the definition of pain today, the recognition of pain as a disease is controversial. Depending on their duration, different types of pain are now classified as chronic pain, and the generally accepted definition is "pain that continues after a normal recovery period."
* The patient's Mini mental test score must be 23 and above. The mini mental state examination is scored on a scale of 0-30 with >25 points interpreted as normal cognitive status.

Exclusion Criteria:

* Those with serious pathological symptoms
* Joint infection
* Cancer
* Rheumatoid arthritis
* Spondyloarthropathy
* Polymyalgia
* Inflammatory arthropathy
* Crystal disease
* Gout
* Those with severe and persistent mental health problems
* Having a diagnosis of dementia
* Those with a terminal illness diagnosis
* Those who have recently experienced trauma or bereavement
* Those who cannot communicate in Turkish
* Those with neurological problems
* Suspected fracture
* Those with joint inflammation
* Those with neuromuscular disease
* Those with systemic disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
The STarT Back Screening Tool | First week
  The STarT Back Screening Tool is a tool designed by Keele University in 2008 to screen prognosis in patients with low back pain in the initial decision-making process.
  It consists of 9 items. Subscale scores range from 0 to 5, and patients with 4 or 5 points are classified in the high-risk subgroup. Scores range from 0-9. Patients with a score of 0-3 are classified as a low-risk subgroup and patients with a score of 4-9 are classified as an intermediate-risk subgroup.
  Cultural adaptation, internal consistency, test repetition and construct validity of the SBST in Turkey were examined in October 2019.

SECONDARY OUTCOMES:
The Roland-Morris Questionnaire (RMDQ) | First week
  The Roland-Morris Questionnaire (RMDQ) was first developed in 1983. It is a self-administered measure of disability in which higher numbers on a 24-point scale reflect greater disability. Its Turkish validity and reliability were demonstrated in 2001. In the questionnaire consisting of 24 sentences about functional deficiencies, patients are asked to answer each sentence as yes if it fits their situation, and no if it doesn't. Calculating yes answers as "1" and no answers as "0", the total score is between 0-24, with a higher score indicating more disability.
Short Form-36 (SF-36) | First week
  Sf-36 was developed and put into use by Rand Corporation in 1992. The scale consists of 36 items and they provide the measurement of 8 dimensions; physical function (10 items), social function (2 items), role limitations due to physical functions (4 items), role limitations due to emotional problems (3 items), mental health (5 items), energy/vitality (4 items), pain (2 items) and general perception of health (5 items) .
  The scale is evaluated considering the last 4 weeks. In order to create the acute form, a form evaluating the last 1 week was also applied. Evaluation 4th and 5th. Apart from the items, Likert type (three-six-point) is made; Items 4 and 5 are answered as yes/no. Instead of giving only a single total score, the scale gives a total score for each subscale separately. Subscales evaluate health between 0 and 100, and 0 includes poor health, while 100 indicates good health
The Tampa Kinesiophobia Scale | First week
  The Tampa Kinesiophobia Scale was originally developed by R.Miller, S.Kopri, and D.Todd in 1991. The Tampa Kinesiophobia Scale (TSK) is a 17-item questionnaire used to assess the subjective rating of kinesiophobia or fear of movement. It was developed to distinguish "non-extreme fear and phobia in patients with chronic musculoskeletal pain". Various studies have found the scale to be a valid and reliable psychometric measure. Initially used to measure fear of movement due to chronic low back pain, TSK was used in different areas including the cervical spine. It is increasingly used for pain related to body parts.TAF is a self-filled questionnaire with a score range of 17 to 68, with higher scores indicating increasing degrees of kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Pamukçu, Principal Investigator — İstinye University
Locations (1):
- İstinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No